CLINICAL TRIAL: NCT01071993
Title: Efficacy Of Statins In The Prevention of Contrast-Induced Nephropathy in Patients With Chronic Renal Insufficiency (SCIN Trial): A Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy of Statins In Prevention of CIN
Acronym: SCIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor can not supply drugs anymore.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15097
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Nephropathy
Keywords: prevention; nephropathy
MeSH Terms: conditions — Kidney Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atorvastatin (Active Comparator)
  Interventions: Drug: atorvastatin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — pre-treatment with placebo (80 mg 12 hours prior to the procedure and 40 mg pre-procedure)
  Arms: placebo
Drug: atorvastatin — pre-treatment with atorvastatin (80 mg 12 hours prior to the procedure and 40 mg pre-procedure)
  Arms: atorvastatin

SUMMARY:
To determine if statin therapy plus intravenous normal saline, in patients with chronic renal insufficiency undergoing angiography, is superior to placebo plus intravenous normal saline therapy in the prevention of CIN.

DETAILED DESCRIPTION:
Due to the conflict in the available data, there are no practice guidelines that are established in order to prevent contrast-induced nephropathy (CIN). Our goal is to determine if statin therapy plus intravenous normal saline, in patients with chronic renal insufficiency undergoing angiography, is superior to placebo plus intravenous normal saline therapy in the prevention of CIN.

ELIGIBILITY:
1. Inclusion Criteria:

   * Adults > 18 years of age
   * undergoing coronary or peripheral angiography with or without intervention
   * Cr > 1.3 mg/dL or GFR < 60 mL/min
2. Exclusion Criteria:

   * end-stage renal disease on dialysis
   * acute renal failure
   * previous iodinated contrast media exposure within 7 days of study entry
   * history of hypersensitivity to statins
   * pregnancy or lactation
   * emergent coronary angiography, ST elevation myocardial infarction (STEMI), or cardiogenic shock
   * prisoners
   * patients already on maximum dose of statins
   * patient receiving N-acetylcysteine or sodium bicarbonate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Abu-Fadel, M.D., Principal Investigator — Oklahoma Univeristy Health Science Center and VA Medical Center
Locations (2):
- United States (2):
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No
No data was collected; therefore, a plan is not applicable.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and signed consent. No drugs were supplied to participants. Study sponsor could not provide study drugs to participants due to cost restraints.
Pre-assignment Details: Prior to assigning participants to specific arms of the protocol, site was informed that the study drug was no longer available.
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants signed consent; however, study was terminated prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint. Development of CIN (Contrast-induced Nephropathy) Defined as a Postprocedure Increase in Serum Creatinine of > 0.5 mg/dL or >25% Increase From Baseline at 24 & at 48 Hours.
Description: Development of CIN (Contrast-induced Nephropathy) Defined as a Postprocedure Increase in Serum Creatinine of > 0.5 mg/dL or >25% Increase From Baseline at 24 & at 48 Hours
Time Frame: 48 hours
Population: Participants signed consent; however, study was terminated prior to randomization
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable/study was terminated prior to randomization.
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study Sponsor no longer supplied study drug/placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No